CLINICAL TRIAL: NCT01499342
Title: Belgian Prospective Multicentre Registry to Evaluate Safety and Performance of the Optimed Stent to Treat Atherosclerotic Lesions in the Superficial Femoral Artery
Brief Title: Belgian Prospective Multicentre Registry to Evaluate Safety and Performance of the Optimed Stent in the Superficial Femoral Artery
Acronym: BOSS
Status: Completed | Type: Observational
Sponsor: be Medical (Industry)
Collaborators: Universitaire Ziekenhuizen KU Leuven (Other); Ziekenhuis Oost-Limburg (Other)
Responsible Party: Sponsor
Other Study IDs: BM/BOSS 02-002
Record Dates: First submitted 2011-04-21; First posted 2011-12-26 (Estimated); Last update posted 2022-08-22 (Actual); Status verified 2014-05

CONDITIONS: Peripheral Arterial Disease
Keywords: Stent; Atherosclerotic occlusive disease; Peripheral arterial disease; Superficial femoral artery; SFA
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Rutherford category 2 - 5

SUMMARY:
This is a Belgian prospective multicentre registry to evaluate safety and performance of the Sinus-Superflex-Visual stent (Optimed) in Superficial Femoral Artery (SFA) atherosclerotic lesions. Target number is 500 patients in approximately 11 centres. Patients will be followed for a period of 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Stenosis (> 75%) or occlusion of the superficial femoral artery (lesion up to 3 cm distal to Hunter's canal and 4 cm proximal to the patella)
* TASC II (2007)type A, B or C lesions
* Target vessel diameter between 4.5 and 7 mm
* Debilitating claudication or critical limb ischemia (Rutherford 2 to 5)
* At least 1 outflow vessel down to the ankle
* Patient is at least 18 years old
* Life expectancy > 2 years
* Patient is compliant with the requested follow-up visits

Exclusion Criteria:

* No informed consent
* Rutherford 6
* TASC II type D lesions
* Patient is not 18 years old
* Patient is pregnant
* Acute ischemia
* Patient is not compliant with the requested follow-up visits
* Unable to cross target lesion with guidewire
* Patient is allergic to nickel-titanium
* Presence of an aneurysm in the SFA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stenosis (> 75%) or occlusion of the superficial femoral artery.
Sampling Method: Non-Probability Sample
Enrollment: 435 (Actual)
Dates: Start 2009-11; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Primary patency | 12, 24 months
  Primary patency rate at 12 and 24 months as determined by Duplex ultrasound, defined as <50% diameter restenosis(systolic velocity ratio no greater than 2.4) at the level of the treated lesion, without occurrence of target lesion revasularization between the index-procedure and the 12 and 24 months follow-up.

SECONDARY OUTCOMES:
Secondary patency | 12 and 24 months
  Patency as defined by absence of >50% restenosis , whether or not after additional intervention to maintain this patency
Target lesion revascularization | 12 and 24 months
  Target lesion revascularisation rate as defined by the number of new revascularizations (endovascular or surgery) carried out due to restenosis or thrombosis at the level of the stented lesion
Target vessel revascularization | 12 and 24 months
  Target vessel revascularization rate as defined by the number of new revascularizations (endovascular or surgery) carried out due to restenosis or a new stenosis in the SFA
Limb-salvage rate | 12 and 24 months
Clinical success rate | 12 and 24 months
  Clinical success rate defined asimprovement in symptoms according to the Rutherford classification by a minimum of 1 class.

CONTACTS AND LOCATIONS:
Overall Officials: Sabrina Houthoofd, MD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven; Herman Schroë, MD, Principal Investigator — Ziekenhuis Oost-Limburg
Locations (2):
- Belgium (2):
  - Ziekenhuis Oost Limburg, Genk, Limburg
  - University Hospital Leuven, Leuven, Vlaams Brabant